CLINICAL TRIAL: NCT01340586
Title: Single-Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Apixaban in Subjects on Hemodialysis
Brief Title: Pharmacokinetics and Pharmacodynamics of Apixaban in Subjects on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CV185-087
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: PHARMACOKINETIC; NOS
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Apixaban (Experimental)
  Interventions: Drug: Apixaban
- Group B: Apixaban (Experimental)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Tablets, Oral, 5 mg, Once, 4 days
  Arms: Group A: Apixaban
Drug: Apixaban — Tablets, Oral, 5 mg, Twice, 15 days
  Arms: Group B: Apixaban

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of a single oral dose of 5 mg Apixaban in subjects with normal renal function and subjects with end stage renal disease (ESRD) maintained with hemodialysis.

DETAILED DESCRIPTION:
Primary Purpose : To provide a clear understanding of the pharmacokinetics of Apixaban in subjects with ESRD and to determine the effect of hemodialysis on Apixaban pharmacokinetics .

ELIGIBILITY:
Inclusion Criteria:

* The signed informed consent form.
* Subjects with normal renal function classified based on calculated creatinine clearance (CLCr) determined by the cockcroft-gault calculation.
* Eligible subjects with ESRD that is maintained with chronic and stable hemodialysis.

Exclusion Criteria:

* Any history of abnormal bleeding or coagulation disorders including those in a first degree relative under 50 years of age.
* History of significant head injury within the last two years.
* Any gastrointestinal surgery that could impact the absorption of study drug.
* Not expected to continue the hemodialysis treatment for the duration of the study.
* INR, PT, or aPTT above the upper limit of normal, unless agreed upon between the investigator and BMS medical monitor.
* History of allergy to Apixaban or Factor Xa inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Orlando, Florida, United States

REFERENCES:
- [Result] Wang X, Tirucherai G, Marbury TC, Wang J, Chang M, Zhang D, Song Y, Pursley J, Boyd RA, Frost C. Pharmacokinetics, pharmacodynamics, and safety of apixaban in subjects with end-stage renal disease on hemodialysis. J Clin Pharmacol. 2016 May;56(5):628-36. doi: 10.1002/jcph.628. Epub 2015 Dec 22. PMID 26331581
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were enrolled in this study. 16 participants were treated and completed the study. Two participants were enrolled but not treated (one withdrew consent, one enrolled as alternate).
Groups:
- Normal Renal Function: Healthy participants with normal renal function (calculated creatinine clearance (ClCr) > 80 mL/min) received a single oral dose of 5 mg apixaban on the morning of Day 1.
- ESRD Maintained With Hemodialysis: Participants with End Stage Renal Disease (ESRD) maintained with hemodialysis received two doses of apixaban separated by a washout period of at least 7 days; one oral dose of 5mg apixaban 2 hours prior to hemodialysis on Day 1 of Period 1, and a second oral dose of 5mg apixaban immediately following the hemodialysis session on Day 1, Period 2.
Period: Overall Study
Arm/Group | Normal Renal Function | ESRD Maintained With Hemodialysis
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | ESRD Maintained With Hemodialysis | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (7.7) | 46.9 (7.9) | 46.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Single 5mg Oral Dose of Apixaban
Description: Maximum observed plasma concentration (Cmax) was measured by plasma concentration of apixaban over time. The geometric means are reported in nanograms per milliliter (ng/mL).
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- ESRD Dose Before Hemodialysis: Participants with ESRD received one oral dose of 5 mg apixaban 2 hours prior to hemodialysis.
- ESRD Dose After Hemodialysis: Participants with ESRD received one oral dose of 5 mg apixaban immediately following the completion of hemodialysis.
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 125.6 (29) | 98.9 (29) | 113.6 (31)
Statistical Analysis 1: Comparison: Normal Renal Function vs ESRD Dose Before Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 0.787, 90% CI 2-sided [0.616 to 1.006]
Statistical Analysis 2: Comparison: Normal Renal Function vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose after hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 0.904, 90% CI 2-sided [0.697 to 1.173]
Statistical Analysis 3: Comparison: ESRD Dose Before Hemodialysis vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over ESRD Dose after hemodialysis; Test type: Superiority or Other; Geometric Mean Ratio = 0.871, 90% CI 2-sided [0.723 to 1.049]

2. Primary Outcome: Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Metabolite BMS-730823
Description: Maximum observed plasma concentration (Cmax) was measured by plasma concentration of BMS-730823 over time. The geometric means are reported in nanograms per milliliter (ng/mL).
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- ESRD Dose Before Hemodialysis: Participants with ESRD received one oral dose of 5 mg apixaban 2 hours prior to hemodialysis on Day 1.
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 10.8 (38) | 15.9 (48) | 20.0 (39)

3. Primary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC(0-T)) of Single 5mg Oral Dose of Apixaban
Description: Area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) was measured by plasma concentration of apixaban over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 1205 (29) | 1430 (41) | 1673 (24)
Statistical Analysis 1: Comparison: Normal Renal Function vs ESRD Dose Before Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 1.187, 90% CI 2-sided [0.907 to 1.553]
Statistical Analysis 2: Comparison: Normal Renal Function vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose after hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 1.389, 90% CI 2-sided [1.097 to 1.758]
Statistical Analysis 3: Comparison: ESRD Dose Before Hemodialysis vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over ESRD Dose after hemodialysis; Test type: Superiority or Other; Geometric Mean Ratio = 0.855, 90% CI 2-sided [0.707 to 1.033]

4. Primary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC(0-T)) of Metabolite BMS-730823
Description: Area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) was measured by plasma concentration of BMS-730823 over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 205 (69) | 746 (56) | 953 (33)

5. Primary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of Single 5mg Oral Dose of Apixaban
Description: The area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) was measured by plasma concentration of apixaban over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 1265 (30) | 1474 (44) | 1717 (24)
Statistical Analysis 1: Comparison: Normal Renal Function vs ESRD Dose Before Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 1.165, 90% CI 2-sided [0.880 to 1.543]
Statistical Analysis 2: Comparison: Normal Renal Function vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose after hemodialysis over Normal Renal Function; Test type: Superiority or Other; Geometric Mean Ratio = 1.357, 90% CI 2-sided [1.066 to 1.728]
Statistical Analysis 3: Comparison: ESRD Dose Before Hemodialysis vs ESRD Dose After Hemodialysis; Geometric Mean Ratio: ESRD Dose before hemodialysis over ESRD Dose after hemodialysis; Test type: Superiority or Other; Geometric Mean Ratio = 0.858, 90% CI 2-sided [0.707 to 1.042]

6. Primary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of BMS-730823
Description: The area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) was measured by plasma concentration of BMS-730823 over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL | NA (NA) — AUC(INF) was excluded due to insufficient profiles | NA (NA) — AUC(INF) was excluded due to insufficient profiles | NA (NA) — AUC(INF) was excluded due to insufficient profiles

7. Primary Outcome: Mean Plasma Terminal Half-life (T-Half) of Single 5mg Oral Dose of Apixaban
Description: Plasma terminal half-life (T-Half) for apixaban was derived from plasma concentrations versus time data. Means were reported in hours.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
hours | 20.0 (14.45) | 12.5 (3.14) | 12.7 (3.40)

8. Primary Outcome: Mean Plasma Terminal Half-life (T-Half) of BMS-730823
Description: Mean plasma terminal half-life (T-Half) for BMS-730823 was derived from plasma concentrations versus time data.
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants with ESRD maintained with hemodialysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
hours | NA (NA) — T-HALF could not be calculated due to a limited number of quantifiable data points on the concentration-time curve

9. Primary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) of a Single 5 mg Oral Dose of Apixaban
Description: Time of maximum observed plasma concentration (Tmax) for apixaban was derived from plasma concentrations versus time data. Medians were reported in hours.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
hours | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 6.0] | 2.00 [2.0 to 6.0]

10. Primary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) of Metabolite BMS-730823
Description: Time of maximum observed plasma concentration (Tmax) for BMS-730823 was derived from plasma concentrations versus time data. Medians were reported in hours.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
hours | 9.00 [6.0 to 12.0] | 15.00 [8.0 to 60.0] | 21.00 [12.0 to 36.0]

11. Primary Outcome: Geometric Mean of Area Under the Plasma Concentration-Time Curve From 2 to 6 Hours (AUC(2-6)) for Apixaban
Description: Area under the plasma concentration-time curve from 2 hours to 6 hours (AUC(2-6) for Apixaban was measured in participants with ESRD during dialysis in Period 1 only. Geometric Means were reported in nanogram hours per milliliter (ng*hr/mL) and were determined from blood samples both entering and exiting the dialyzer.
Time Frame: 2 to 6 hours post-dose
Population: All participants with ESRD maintained with hemodialysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
ng*hr/mL
  Blood entering dialyzer | 309 (29)
  Blood exiting dialyzer | 312 (28)

12. Primary Outcome: Geometric Mean of Area Under the Plasma Concentration-Time Curve From 2 to 6 Hours (AUC(2-6)) for BMS-730823
Description: Area under the plasma concentration-time curve from 2 hours to 6 hours (AUC(2-6) for BMS-730823 was measured in participants with ESRD during dialysis in Period 1 only. Geometric Means were reported in nanogram hours per milliliter (ng*hr/mL) and were determined from blood samples both entering and exiting the dialyzer.
Time Frame: 2 to 6 hours post-dose
Population: All participants with ESRD maintained with hemodialysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
ng*hr/mL
  Blood entering dialyzer | 15.0 (102)
  Blood exiting dialyzer | 17.7 (96)

13. Primary Outcome: Mean Percent Dose of Apixaban Recovered in Urine (%UR)
Description: The percent dose recovered in urine was calculated by dividing the cumulative amount of unchanged apixaban excreted in urine from the time of dose up to 72 hours post-dose by the apixaban dose administered.
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: percent of dose recovered in urine
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
percent of dose recovered in urine | 18.397 (8.5545) | 0.145 (0.0881) | 0.181 (0.1391)

14. Primary Outcome: Mean Percent Dose of Apixaban Recovered in Dialysate (%DR)
Description: Percent dose of Apixaban recovered in dialysate (%DR) was calculated by dividing the cumulative amount of apixaban excreted in each dialysate collection over 2-6 hours (DR(2-6)) by the apixaban dose. %DR was recorded only in period 1.
Time Frame: 2 to 6 hours post-dose
Population: All treated participants with ESRD maintained with hemodialysis
Measure: Mean (Standard Deviation); unit: percent of dose recovered in dialysate
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
percent of dose recovered in dialysate | 6.68 (1.408)

15. Primary Outcome: Mean Renal Clearance (CLR) of Apixaban
Description: Renal clearance (CLR) was calculated by dividing the cumulative amount of apixaban excreted in urine by the respective cumulative plasma AUC over the same urine collection interval. Geometric means were reported in milliliters per minute (mL/min).
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
mL/min | 11.263 (44) | 0.020 (70) | 0.020 (80)

16. Primary Outcome: Mean Renal Clearance (CLR) of BMS-730823
Description: Renal clearance (CLR) was calculated by dividing the cumulative amount of BMS-730823 excreted in urine by the respective cumulative plasma AUC over the same urine collection interval. Geometric means were reported in milliliters per minute (mL/min).
Time Frame: 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
mL/min | 6.36 (62) | NA (NA) — Parameters cannot be estimated for ESRD group due to functional anuria or below Lower Level of Quantitation (LLOQ) | NA (NA) — Parameters cannot be estimated for ESRD group due to functional anuria or below Lower Level of Quantitation (LLOQ)

17. Primary Outcome: Mean Hemodialysis Clearance (CLD) of Apixaban
Description: Hemodialysis clearance (CLD) was calculated by dividing the cumulative amount of apixaban excreted in dialysate by the respective cumulative plasma AUC over the same dialysate collection interval (AUC(2-6) entering). CLD measurements occurred only in period 1. Geometric means were reported in milliliters per minute (mL/min).
Time Frame: 2 to 6 hours post-dose
Population: All treated participants with ESRD maintained with hemodialysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
mL/min | 17.7 (19)

18. Primary Outcome: Mean Hemodialysis Clearance (CLD) of BMS-730823
Description: Hemodialysis clearance (CLD) was calculated by dividing the cumulative amount of BMS-730823 excreted in dialysate by the respective cumulative plasma AUC over the same dialysate collection interval (AUC(2-6) entering). CLD measurements occurred only in period 1. Geometric means were reported in milliliters per minute (mL/min).
Time Frame: 2 to 6 hours post-dose
Population: All participants with ESRD maintained with hemodialysis
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
mL/min | NA (NA) — CLD for BMS-730823 was not determined since concentration in all dialysate samples were below Lower Level of Quantitation (LLOQ)

19. Primary Outcome: Percentage of Apixaban Extracted During Hemodialysis
Description: The percentage of apixaban extracted during hemodialysis (extraction ratio) was calculated using the formula [plasma AUC(2-6) exiting - AUC(2-6) entering] / [AUC(2-6) entering] and converted to a percentage. The extraction ratio was measured in period 1 only, and was reported as a percentage.
Time Frame: 2 to 6 hours post-dose
Population: All treated participants with ESRD maintained with hemodialysis
Measure: Mean (Standard Deviation); unit: percentage of apixaban extracted
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
percentage of apixaban extracted | -1.1 (5.65)

20. Primary Outcome: Percentage of BMS-730823 Extracted During Hemodialysis
Description: The percentage of BMS-730823 extracted during hemodialysis (extraction ratio) was calculated using the formula [plasma AUC(2-6)exiting - AUC(2-6)entering] / [AUC(2-6) entering] and converted to a percentage. The extraction ratio was measured in period 1 only, and was reported as a percentage.
Time Frame: 2 to 6 hours post-dose
Population: All treated participants with ESRD maintained with hemodialysis
Measure: Mean (Standard Deviation); unit: percentage of BMS-730823 extracted
Arm/Group | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8
percentage of BMS-730823 extracted | -19.9 (25.32)

21. Secondary Outcome: Mean Maximum Percent Change From Baseline International Normalized Ratio (INR) Following a Single 5 mg Oral Dose of Apixaban
Description: The mean maximum percent change in baseline for INR was reported for each arm. Baseline measurements were assessed up to 24 hours prior to Day 1 dosing.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: maximum percent change from baseline
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
maximum percent change from baseline | 31.5 (56.59) | 16.6 (10.60) | 16.8 (7.15)

22. Secondary Outcome: Mean Maximum Percent Change From Baseline Prothrombin Time (PT) Following a Single 5 mg Oral Dose of Apixaban
Description: The mean maximum percent change in Prothrombin Time (PT) from baseline was reported for all treated participants. Baseline measurements were assessed up to 24 hours prior to Day 1 dosing.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: maximum percent change from baseline
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
maximum percent change from baseline | 32.4 (58.31) | 16.9 (10.98) | 17.4 (7.28)

23. Secondary Outcome: Mean Maximum Percent Change From Baseline Activated Partial Thromboplastin Time (aPTT) Following a Single Oral Dose of 5 mg Apixaban
Description: The mean maximum percent change in Activated Partial Thromboplastin Time (aPTT) from baseline was reported for all treated participants. Baseline measurements were assessed up to 24 hours prior to Day 1 dosing.
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: maximum percent change from baseline
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
maximum percent change from baseline | 19.9 (20.40) | 7.0 (9.62) | 23.0 (14.81)

24. Secondary Outcome: Mean Peak Anti-FXa Activity Following a Single Oral Dose of 5 mg Apixaban
Description: Anti-FXa activity was assessed from an activity-time profile for doses both before and after hemodialysis. Maximal means were reported in International Units per milliliter (IU/mL).
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Number analyzed (Participants) | 8 | 8 | 8
IU/mL | 1.47 (0.659) | 1.03 (0.491) | 1.29 (0.579)

25. Other Pre Specified Outcome: Number of Participants With Laboratory Marked Abnormalities
Description: ULN=Upper Limit of Normal, LLN=Lower Limit of Normal, Pre-Rx= Baseline value. BUN=Blood Urea Nitrogen (mmol/L=millimoles per Liter): High if BUN > 1.1*ULN (if Pre-Rx>ULN: >1.25*Pre-Rx).
  Platelet count (*10^9 cell/L): Low if Platelet Count < 0.85*LLN (if Pre-Rx<LLN: <0.85*Pre-Rx).
  Creatine (umol/L=micromoles per Liter): High if Creatine > 1.5*ULN (if Pre-Rx>ULN: >1.33*Pre-Rx).
  Calcium, Total (mmol/L): High if Calcium > 1.5*ULN (if Pre-Rx>ULN: >1.33*Pre-Rx).
  Potassium, serum (mmol/L): High if Potassium > 1.1*ULN (if Pre-Rx>ULN: >1.1*Pre-Rx; if Pre-Rx<LLN: >ULN).
  Phosphorus, Inorganic (mmol/L): Low if Phosphate < 0.85*LLN (if Pre-Rx>ULN: <LLN).
  Lactate dehydrogenase (U/L=Units per Liter): High if Lactate Dehydrogenase > 1.25*ULN (if Pre-Rx>ULN: >1.5*Pre-Rx).
Time Frame: From 24 hours pre-dose to 72 hours post-dose
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8 | 8
participants
  BUN | 0 | 4
  Platelet count | 0 | 1
  Creatine | 0 | 1
  Potassium | 0 | 1
  Phosphorus | 0 | 1
  Lactate dehydrogenase | 0 | 1

26. Other Pre Specified Outcome: Number of Participants Who Died or Experienced Serious Adverse Events (SAEs) or Adverse Events Leading to Discontinuation
Description: The number of participants who died or experienced SAEs or AEs leading to discontinuation was reported for each arm.
  AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling.
Time Frame: From Day 1 to 30 days post study discontinuation
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | ESRD Maintained With Hemodialysis
Number analyzed (Participants) | 8 | 8
participants
  Deaths | 0 | 0
  SAEs | 0 | 0
  AEs leading to discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 until 30 days post discontinuation, up to September 2011 (approximately 3 months)
Description: Study initiated: June 2011
  Study completed: September 2011
  Participants underwent regular laboratory testing and investigator assessment as outlined in the study protocol.
Arm/Group | Normal Renal Function | ESRD Dose Before Hemodialysis | ESRD Dose After Hemodialysis
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 2/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | ESRD Dose Before Hemodialysis (N=8) | ESRD Dose After Hemodialysis (N=8)
Headache (Nervous system disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.